CLINICAL TRIAL: NCT07299214
Title: The Effect of Music During Non-Stress Testing on Women's Comfort, Vital Signs and Anxiety: A Randomized Controlled Study
Brief Title: Music During Non-Stress Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, GAMZE GOKE ARSLAN, Asistant Professor, Department of Nursing, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMBU-NST-2025-01; 2169 (Ethics decision number) (Other: Non-Interventional Clinical Research Ethics Committee of the Republic of Türkiye Izmir Bakırçay University)
Record Dates: First submitted 2025-11-23; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pregnant Women
Keywords: non-stress test; music; comfort; vital signs; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Simple randomization method was used in this study. Pregnant women who met the study criteria were randomly assigned to the music or control group with equal probability, independently of any previous assignments, on the day they came to the hospital for their physical examination. The total number of pregnant women determined by the G*Power analysis was entered into the program at ''https://www.randomizer.org," and randomization was conducted using the program. The assignment of the groups was performed on the computer, and the pregnant women were randomly assigned to the music and control groups. The data of the study were collected from the pregnant women using the face-to-face interview technique at the NST outpatient clinic on the days and hours when the researcher was present in the hospital.
Who Masked: Participant
Masking Description: The participating pregnant women were not informed of the group they belonged to. Since only the researcher knew the participants' groups, single-blindness was achieved in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): After the pregnant women were positioned, while the NST procedure was implemented they listened to music for 20-30 minutes. The pregnant women listened to the music on an MP3 player during the application. The duration of the music recorded on the MP3 player was 30 minutes. The music played to the pregnant women was selected by the researchers in accordance with the definition of relaxing music made in the literature. Before the music selection, the researchers communicated with the TÜMATA (Turkish acronym for the "Research and Promotion of Turkish Music Association). After the meeting held with the association, it was decided to use the 'Acemaşiran' (a musical mode in traditional Turkish music). In the study, music prepared by the TÜMATA in the Acemaşiran mode was played. It is stated that Acemaşiran mode helps balance the body, helps the listener relax, facilitates birth, helps correct the wrong position of the fetus in the womb, and has a pain and spasm relieving effect
  Interventions: Other: Music intervention
- Control Group (No Intervention): Pregnant women were not subjected to any intervention during the NST procedure.

INTERVENTIONS:
Other: Music intervention — The music played to the pregnant women was selected by the researchers in accordance with the definition of relaxing music made in the literature. Before the music selection, the researchers communicated with the TÜMATA (Turkish acronym for the "Research and Promotion of Turkish Music Association). After the meeting held with the association, it was decided to use the 'Acemaşiran' (a musical mode in traditional Turkish music). In the study, music prepared by the TÜMATA in the Acemaşiran mode was played. It is stated that Acemaşiran mode helps balance the body, helps the listener relax, facilitates birth, helps correct the wrong position of the fetus in the womb, and has a pain and spasm relieving effect.
  Arms: Music Group

SUMMARY:
Music has direct and indirect positive effects on the mother and fetus during pregnancy and perinatal period. This study was aimed at investigating effects of music played during the Non-Stress Test (NST) procedure on the mother's comfort, vital signs and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years
* Completion of at least the 32nd week of gestation
* No pregnancy-related risk factors (e.g., premature rupture of membranes, preeclampsia, gestational diabetes)
* No multiple pregnancy
* Normal blood pressure levels (not ≤80/60 mmHg and not ≥140/90 mmHg)
* Having eaten at least two hours before the NST procedure
* No smoking or alcohol consumption for at least two hours before the NST procedure
* Ability to communicate effectively
* No hearing impairment
* Voluntary participation in the study

Exclusion Criteria:

* Pregnant women with fetal distress
* Cases for whom the physician considered emergency intervention necessary
* Individuals with an impaired NST requiring immediate intervention
* Individuals with a diagnosed psychiatric disorder
* Individuals with hearing impairment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participation in the study was restricted based on biological sex. Because the study included pregnant women, biologically female individuals were eligible to participate.
Enrollment: 173 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
During Non-Stress Testing on Women's Comfort Level | Pre-test: Before NST application Post-test: After NST application (Approximately 20-30 minutes after the NST session begins)
  Prenatal Comfort Scale (PCS) was used to determine women's comfort level. The short version of the PCS consists of 15 items. Response given to the items are rated on a six-point Likert type scale ranging from 0 to 5 (0 = Strongly disagree, 1 = Disagree, 2 = Undecided, 3 = Somewhat agree, 4 = Agree, 5 = Strongly agree). The minimum and maximum possible scores that can be obtained from the PCS are 0 and 75, respectively. The higher the score is the higher the comfort level is.
During Non-Stress Testing on Women's Systolic Blood Pressure Level | Pre-test: Before NST application Post-test: After NST application (Approximately 20-30 minutes after the NST session begins)
  The women's systolic blood pressure levels were measured with a calibrated electronic sphygmomanometer. Blood pressure levels are expressed in millimeters of mercury (mmHg).
During Non-Stress Testing on Women's Diastolic Blood Pressure Level | Pre-test: Before NST application Post-test: After NST application (Approximately 20-30 minutes after the NST session begins)
  The women's diastolic blood pressure levels were measured with a calibrated electronic sphygmomanometer. Blood pressure levels are expressed in millimeters of mercury (mmHg).
During Non-Stress Testing on Women's Diastolic Heart Rate Level | Pre-test: Before NST application Post-test: After NST application (Approximately 20-30 minutes after the NST session begins)
  Heart rate level was determined electronically. Heart rate level was recorded in beats per minute (bpm).
During Non-Stress Testing on Women's Anxiety Level | Pre-test: Before NST application Post-test: After NST application (Approximately 20-30 minutes after the NST session begins)
  State Anxiety Scale (SAS) was used to determine the anxiety level. The scale is a 4-point Likert type, "not at all" (1), "somewhat" (2), "moderately" (3), "very much" (4). The scale consists of 20 items and items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reverse scored. To calculate the total score of the SAS, the total score of the reversed items is subtracted from the total score of the non-reversed items. Then, 50 points, which is the constant value of the state anxiety scale, are added to this score. The result is the score for the overall SAS. The total score varies between 20 and 80. The higher the score is the higher the level of the anxiety is. While a score ranging between 0 and 19 indicates "no anxiety", a score ranging between 20 and 39 indicates mild anxiety, a score ranging between 40 and 59 indicates moderate anxiety, a score ranging between 60 and 79 indicates severe anxiety, and a score of 80 indicates very severe anxiety (Panic).

CONTACTS AND LOCATIONS:
Locations (1):
- University District, 2076 Street, No: 11, Karaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT07299214/Prot_SAP_ICF_000.pdf